CLINICAL TRIAL: NCT06964698
Title: Erector Spinae Plane Block Versus Paravertebral Block for Post-Thoracotomy Pain Syndrome in Thoracotomy Patients; A Prospective Observational Study
Brief Title: Optimizing Post-Thoracotomy Pain Management: Comparing Erector Spinae vs. Paravertebral Block in Thoracotomy Patients
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Ozal Adiyeke, specialist, MD, Başakşehir Çam & Sakura City Hospital
Other Study IDs: KAEK.2022.05.155
Record Dates: First submitted 2025-04-02; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Lung Diseases; Lung Cancers
Keywords: thoracotomy; erector spinae plane block; paravertebral block; post-operative pain syndrome
MeSH Terms: conditions — Lung Diseases; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paravertebral Block (PVB): Includes patients with paravertebral block as analgesic For the PVB, the patient was seated, and a 22G block needle was inserted into the paravertebral space at the T5 level under ultrasound guidance. The T5 level was selected to provide direct analgesia to the thoracic paravertebral space, which is known to block multiple thoracic nerves. After negative aspiration, 1 mL of saline was injected to confirm correct needle placement, and 20 mL of 0.375% bupivacaine was administered following hydrodissection.
- Erector Spinae Plane Block (ESPB): Includes patients with Erector Spinae Plane Block as analgesic. For ESPB, the patient was positioned in a seated posture, and under sterile conditions, a 22G, 80 mm Stimuplex® D block needle (B. Braun, Melsungen, Germany) was inserted between the T6 and T7 transverse processes and the erector spinae muscle via ultrasound guidance (Fujifilm Arietta 65, Tokyo, Japan). The T6-T7 level was chosen on the basis of its proximity to the thoracic surgical site, allowing for optimal coverage of the thoracic dermatomes. Following negative aspiration, 1 mL of saline was injected via hydrodissection to confirm correct needle placement, and 20 mL of 0.375% bupivacaine was administered.

SUMMARY:
This prospective, observational study included ASA class II-III patients aged 18-70 years who underwent elective unilateral lobectomy via a thoracotomy. The study was conducted at Başakşehir Çam and Sakura City Hospital, following approval from the hospital's ethics committee on May 20, 2022 (protocol number: KAEK.2022.05.155). Patients were randomized into two groups based on the type of preoperative block administered: ESPB (n = 30) and PVB (n = 30). Intravenous patient-controlled analgesia was provided for 24 hours postoperatively. Resting NRS and Prince Henry Hospital Pain Scale (PHHPS) scores were evaluated at 0, 2, 6, 12, and 24 hours after surgery. Pain levels were further assessed via telephone interviews using the NRS at 2 weeks and 2 months postoperatively.

DETAILED DESCRIPTION:
Study Design and Ethics Approval It was conducted as a prospective, observational trial at the Basaksehir Cam and Sakura City Hospital, after approval had been obtained from the ethics committee of the Basaksehir Cam and Sakura City Hospital on May 20,2022, (protocol number: KAEK.2022.05.155). Our study recognises the Declaration of Helsinki as a statement of ethical principles for medical research involving human participants.

Patient Population and Randomization Adult patients aged 18-70 years who underwent unilateral lobectomy via a thoracotomy approach under elective conditions between June 1, 2022, and December 1, 2022, were included in the study. Informed consent was obtained from all patients prior to enrollment. The inclusion criteria were as follows: patients classified as ASA II-III, no history of previous thoracotomy, no chronic pain or analgesic dependence, and adequate preoperative cooperation. The exclusion criteria included patients with known drug allergies, chronic analgesic use, or preexisting neuropathic conditions.

Randomization was performed via a computer-generated sequence to ensure the true random allocation of patients into either the ESPB or the PVB group. The sequence was concealed via sealed opaque envelopes, which were opened by the attending anesthesiologist just before block administration. No stratification was applied; however, group assignment was conducted to ensure an equal distribution of patients by sex, age, and ASA status. The anesthesiologist monitoring postoperative pain was blinded to the type of block administered.

Preoperative anaesthesia preparation and block protocols All patients received standard ASA monitoring, including invasive blood pressure measurement. All blocks were performed by the same anesthesiologist (O.A.), who had more than 7 years of experience in ultrasound-guided regional anesthesia.

Erector Spinae Plane Block (ESPB) Protocol For ESPB, the patient was positioned in a seated posture, and under sterile conditions, a 22G, 80 mm Stimuplex® D block needle (B. Braun, Melsungen, Germany) was inserted between the T6 and T7 transverse processes and the erector spinae muscle via ultrasound guidance (Fujifilm Arietta 65, Tokyo, Japan). The T6-T7 level was chosen on the basis of its proximity to the thoracic surgical site, allowing for optimal coverage of the thoracic dermatomes. Following negative aspiration, 1 mL of saline was injected via hydrodissection to confirm correct needle placement, and 20 mL of 0.375% bupivacaine was administered.

Paravertebral block (PVB) protocol For the PVB, the patient was seated, and a 22G block needle was inserted into the paravertebral space at the T5 level under ultrasound guidance. The T5 level was selected to provide direct analgesia to the thoracic paravertebral space, which is known to block multiple thoracic nerves. After negative aspiration, 1 mL of saline was injected to confirm correct needle placement, and 20 mL of 0.375% bupivacaine was administered following hydrodissection.

Anaesthesia Protocol Premedication was achieved with 2 mg intravenous midazolam, which was administered prior to the block performance. General anaesthesia induction was achieved with 2 mcg/kg fentanyl and 1.5-3 mg/kg propofol, with a target bispectral index (BIS) between 40 and 60. Neuromuscular blockade was induced via 0.6 mg/kg rocuronium, and maintenance of anaesthesia was achieved via sevoflurane (1%-2%) and remifentanil (0.05--0.2 mcg/kg/min) in a 50% oxygen/air mixture. All patients underwent orotracheal intubation with a double-lumen tube appropriate for their body height and surgical side, and mechanical ventilation parameters were standardized across all patients. A standard posterolateral thoracotomy was performed through the fifth intercostal space to provide surgical access. For optimal postoperative drainage and lung re-expansion, a 28 Fr chest tube was inserted through the sixth intercostal space, one level below the thoracotomy incision. All operations were carried out by the same team.

At the conclusion of the surgery, patients were administered 1 g of paracetamol and 100 mg of tramadol intravenously, followed by decurarization with 2-4 mg/kg sugammadex. A patient-controlled analgesia (PCA) device (BodyGuard 595) with a basal infusion of 2.5 mL/h of tramadol (500 mg tramadol in 125 mL of 0.9% NaCl) was used for postoperative analgesia (intermittent bolus dose of 5 mL - lock time 30 min). Morphine (0.1 mg/kg) was used as a rescue analgesic if the NRS score exceeded 4 out of 10.

Outcome Measurements The primary outcome was postoperative pain, which was assessed via the NRS and the Prince Henry Hospital Pain Scale (PHHPS) at 0, 2, 6, 12, and 24 hours postoperatively. Pain levels were also assessed at 2 weeks and 2 months postoperatively, with phone calls for follow-up. Although phone assessments may introduce bias due to the subjective nature of self-reported pain levels, this method was chosen to maintain follow-up consistency across all patients. To mitigate this limitation, the same standardized questionnaire was used for all phone assessments, and patients were instructed to report their pain levels accurately.

The secondary outcomes included the incidence of PTPS at 2 months, the total consumption of opioids via the PCA device, the number of requests for rescue analgesia, and the incidence of complications such as hematoma, pneumothorax, or nerve damage. Additionally, demographic characteristics, intraoperative hemodynamic data, and surgical duration were recorded.

The secondary outcomes included the incidence of PTPS at 2 months; the total consumption of opioids via the PCA device at 24 hours postoperatively; the number of requests for rescue analgesia within the first 24 hours postoperatively; and the incidence of complications such as hematoma, pneumothorax, or nerve damage. Hemodynamic variables were assessed with measurements taken at the following predefined times: preoperatively, end of induction, time of skin incision, 30th, 60th, 90th and 120th minute of block and end of surgery. Additionally, demographic characteristics, intraoperative hemodynamic data, and surgical duration were recorded.

Statistical analysis A power analysis was conducted to determine the required sample size, with an alpha of 0.05 and beta of 0.1, expecting a minimum 3 mg difference in 24-hour opioid consumption between the groups (doi: 10.7759/cureus.59459). Based on an estimated effect size of Cohen's d ≈ 0.9, a minimum of 60 patients (30 per group) were included to achieve a power of 90%. A total of 64 patients were enrolled to account for potential attrition. The data were analysed via SPSS (Mac OS, version 27.0). The normality of the data was assessed with the Kolmogorov-Smirnov test. Normally distributed data were analyzed using independent t-tests, while non-normally distributed data were analyzed with the Mann-Whitney U test. Categorical variables were compared using chi-square or Fisher's exact tests. Continuous variables are presented as the means ± standard deviations, and categorical variables are presented as frequencies and percentages. Statistical significance was determined by p values < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients were planned to elective thoracotomy
* Patients classified as ASA II-III,
* No history of previous thoracotomy,
* No chronic pain or analgesic dependence,
* Adequate preoperative cooperation.

Exclusion Criteria:

* Known drug allergies
* Chronic analgesic use
* Preexisting neuropathic conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18-70 years who underwent unilateral lobectomy via a thoracotomy approach under elective conditions
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
The numeric rating scale (NRS) | The numeric rating scale (NRS) was assessed at 0, 2, 6, 12 and 24 hours, 2 weeks and 2 months postoperatively,
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable.
The Prince Henry Hospital Pain Scale (PHHPS) | The Prince Henry Hospital Pain Scale (PHHPS) was assessed at 0, 2, 6, 12 and 24 hours, 2 weeks and 2 months postoperatively,
  The Prince Henry Hospital Pain Scale is a pain screening tool at physical activity. Pain is estimated during elementary physical activity: 0 - no pain, cough, 1 - pain when coughing, lack during deep breathing, 2 - pain during deep breathing, lack of rest, 3 - slight pain at rest, 4 - severe pain at rest.

SECONDARY OUTCOMES:
The incidence of post-thoracotomy pain syndrome | The incidence of post-thoracotomy pain syndrome was assessed at 2 months postoperatively.
  The incidence of post-thoracotomy pain syndrome is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable.
The number of request of opioids | The number of request of opioids was assessed at 24 hours postoperatively.
  The number of request of opioids via the PCA device was accessed.
The incidence of complications | The incidence of complications was assessed at 24 hours postoperatively.
  Complications such as hematoma, pneumothorax, or nerve damage was accessed.
The total consumption of opioids | The total consumption of opioids was assessed at 24 hours postoperatively.
  The total consumption of opioids via the PCA device was accessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam Ve Sakura Şehir Hastanesi, Istanbul, Basaksehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol